CLINICAL TRIAL: NCT06787521
Title: PEAICE: Patient Empowerment and Agency Through Intrapartum Counseling and Education: a Randomized Controlled Study
Brief Title: Patient Empowerment and Agency Through Intrapartum Counseling and Education
Acronym: PEAICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Fei Cai, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OHSU IRB 28141
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related
Keywords: Intrapartum; Labor Agency

STUDY DESIGN:
Intervention Model Description: 1:1 randomization will be done using REDCap.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants will receive an evidence-based labor guide at the time of admission for scheduled induction of labor
  Interventions: Other: evidence-based labor guide
- Control Group (No Intervention): Participants will receive the standard of care in-person counseling regarding options for labor interventions.

INTERVENTIONS:
Other: evidence-based labor guide — Participants will be provided with written education about potential complications and interventions. Information will be provided at the time of admission for labor induction.
  Arms: Experimental Group

SUMMARY:
A single-blind randomized controlled trial to study the effects of a labor guide on perceived control in labor. The experimental arm will receive an evidence-based labor guide at the time of admission for scheduled induction of labor. The control arm will receive the standard of care in-person counseling regarding options for labor interventions

DETAILED DESCRIPTION:
Participants will be randomized to receive an evidence-based labor guide at the time of admission for scheduled induction of labor, or the standard of care. Following delivery, patients will be surveyed about their labor experience. Chart review will be done to collect data on obstetric interventions and outcomes and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Singleton pregnancy
* English-speaking
* Undergoing induction of labor for a medical or elective indication
* Reached at least 36 weeks 0 days gestation
* Willing and able to sign a consent form
* Delivering at OHSU

Exclusion Criteria:

* Undergoing induction termination
* Fetal complications such as multiple gestation, major fetal anomalies, fetal demise
* Decisionally-impaired adults
* Minors

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Labor Agentry Scale-10 (LAS-10) | 1-7 days following delivery
  A validated questionnaire that measures patient-perceived control during labor

SECONDARY OUTCOMES:
Labor Interventions | During labor
  Whether patients received labor interventions including Pitocin, misoprostol, cook balloon, intra-uterine pressure catheter, manual rotation
Maternal hyper/hypotension | During induction of labor
  Whether the patient experience hypertension or hypotension
Intrapartum blood loss | Labor and delivery
  The amount of blood loss a patient experienced during delivery
Cesarean section | Delivery
  Whether a patient requires a cesarean delivery
Time to delivery | Admission for induction to delivery
  The duration from admission for induction to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Fei Cai, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No